CLINICAL TRIAL: NCT06601959
Title: Study Protocol for Measuring Energy Needs and Nutritional Status of Adolescent Girls in Abia State, Nigeria: The Nutrition and Adolescence in Rural Nigeria (NARN'ia) Study
Brief Title: Energy Needs and Nutritional Status of Adolescent Girls
Acronym: NARNia
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00114378; INV-061141 (Other Grant/Funding Number: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-10

CONDITIONS: Nutrition; Energy Requirement
Keywords: Nutrition; Energy requirements; female adolescents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescent female students: Adolescent female students from elementary to secondary schools in the Ikwuano Local Government Area of Abia State, Nigeria

SUMMARY:
The purpose of this study is to investigate the energy needs and nutritional status of adolescent girls in Abia State, Nigeria

DETAILED DESCRIPTION:
Adolescents in low and middle-income countries encounter numerous nutritional challenges, including undernutrition, micronutrient deficiencies, poor dietary habits, and food insecurity. These issues significantly impact their growth, development, and long-term health. Despite their increased vulnerability, this demographic is often overlooked in nutritional program planning and implementation. This neglect is due to a lack of accurate data, inadequate delivery platforms for interventions, and underdeveloped policies and programs.

The Nutrition and Adolescence in Rural Nigeria (NARN'ia) study aims to address this gap through a comprehensive assessment of energy requirements in adolescent girls (N=50; ages 10 - 19 years) in Nigeria. NARN'ia will integrate dietary assessments using the 24-hour recall method (INDDEX24 app); physical activity levels using accelerometry; anthropometric evaluations of body composition, and the doubly labeled water method for assessing both body composition and total daily energy expenditure.

This study will provide evidence-based data essential for formulating appropriate nutritional guidelines for adolescent girls in Nigeria. Furthermore, this research initiative will establish a foundational framework for future studies on energy requirements in Nigeria and other low and middle-income countries.

ELIGIBILITY:
Inclusion Criteria:

* female students
* 10 and 19 years old
* provides verbal assent and has parental consent

Exclusion Criteria:

* physical disabilities
* illnesses during the study period
* students attending boarding schools

Ages: 10 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Cisgender adolescent girls
Study Population: The NARN'ia study will be conducted in Ikwuano Local Government Area of Abia State, located in southeast Nigeria. Ikwuano is a rural region primarily inhabited by crop farmers and traders from the Igbo ethnic group. Participants (n=50) will be recruited from four secondary schools in Ikwuano.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Total Energy Expenditure measured with Doubly Labeled Water (DLW) | 10 days from enrollment
  The rate of elimination of hydrogen and oxygen isotopes from the DLW through urine will be used to estimate TEE in kilocalories per day (kcal/day).
Physical Activity Levels using a wrist-worn accelerometer | 10 days from enrollment
  Physical activity levels will be categorized under light, moderate, and vigorous and will be expressed as accelerations over each day.
  Light Physical Activity: Acceleration: 0.05 g to 0.1 g Moderate Physical Activity:Acceleration: 0.1 g to 0.3 g Vigorous Physical Activity:Acceleration: ≥ 0.3 g
  This will be reported as the number of participants at each physical activity level.
Dietary Intake using the INDDEX24 app - total energy (kcal/day) content | 10 days from enrollment
  The INDDEX24 dietary recall app will be used to capture detailed information on all foods and beverages consumed during the recall period. Nutritional intake will be analyzed for total energy (kcal/day).
Dietary Intake using the INDDEX24 app - macronutrient content | 10 days from enrollment
  The INDDEX24 app will be used to assess the macronutrient consumed by each individual per day over the course of the enrollment period.
Dietary Intake using the INDDEX24 app - micronutrient content | 10 days from enrollment
  The INDDEX24 app will be used to access the micronutrient content of the diets of the participants for the duration of enrollment.
Body composition - BMI | 10 days from enrollment
  Body composition will be assessed by recording the heights and weights of the participants with a tape measure and body scale respectively to calculate their body mass indices (BMI) in kg/m^2
Body composition - skinfold thickness (biceps) | 10 days from enrollment
  Body composition will be assessed by recording biceps skinfold thickness of the participants using skinfold calipers in mm.
Body composition - skinfold thickness (triceps) | 10 days from enrollment
  Body composition will be assessed by recording triceps skinfold thickness of the participants using skinfold calipers in mm.
Body composition - skinfold thickness (subscapular) | 10 days from enrollment
  Body composition will be assessed by recording subscapular skinfold thickness of the participants using skinfold calipers in mm.
Body composition - skinfold thickness (suprailiac) | 10 days from enrollment
  Body composition will be assessed by recording suprailiac skinfold thickness of the participants using skinfold calipers in mm.
Body composition - waist circumference | 10 days from enrollment
  Body composition will be assessed by recording the waist circumference of the participants using a tape measure in cm.
Body composition - hip circumference | 10 days from enrollment
  Body composition will be assessed by recording the hip circumference of the participants using a tape measure in cm.

CONTACTS AND LOCATIONS:
Overall Officials: Herman Pontzer, Principal Investigator — Duke University Evolutionary Anthropology
Locations (2):
- Duke University Evolutionary Anthropology, Durham, North Carolina, United States
- Michael Okpara Universty of Agriculture, Umudike, Abia State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data (IPD) from this study, including measurements of body composition (height, waist circumference, hip circumference, skinfold thickness, body weight, and bioelectrical impedance results), physical activity levels (accelerometry data), total energy expenditure (DLW data), and dietary intake (INDDEX24 app data), will be made available upon reasonable request. All personal identifiers will be removed to ensure participants' privacy and confidentiality.
Supporting Information: Study Protocol
Time Frame: Beginning 1 year after publication with no end date
Access Criteria: Researchers interested in accessing the anonymized dataset must submit a formal request outlining the intended use of the data. Requests will be reviewed by the study's principal investigator to ensure appropriate use. Data access will be granted through a secure data-sharing platform, and users will be required to sign a data-sharing agreement to ensure that the data is used exclusively for research purposes and in line with ethical guidelines. The shared dataset will include:
  Body Composition Data: Height, waist and hip circumference, skinfold thickness, body weight, and bioelectrical impedance results.
  Accelerometry Data: Physical activity levels, including step counts, intensity (light, moderate, vigorous), and sedentary behavior over the study period.
  DLW Data: Total energy expenditure (TEE) estimates derived from the doubly labeled water method.
  Dietary Intake Data: Nutritional intake recorded via the INDDEX24 app, including energy and macronutrient intake

REFERENCES:
- [Background] Fomon SJ, Haschke F, Ziegler EE, Nelson SE. Body composition of reference children from birth to age 10 years. Am J Clin Nutr. 1982 May;35(5 Suppl):1169-75. doi: 10.1093/ajcn/35.5.1169. No abstract available. PMID 7081099
- [Background] Oyeyemi AL, Umar M, Oguche F, Aliyu SU, Oyeyemi AY. Accelerometer-determined physical activity and its comparison with the International Physical Activity Questionnaire in a sample of Nigerian adults. PLoS One. 2014 Jan 28;9(1):e87233. doi: 10.1371/journal.pone.0087233. eCollection 2014. PMID 24489876
- [Background] Boreham C, Riddoch C. The physical activity, fitness and health of children. J Sports Sci. 2001 Dec;19(12):915-29. doi: 10.1080/026404101317108426. PMID 11820686
- [Background] Coates J, Bell W, Bakun P, Adams KP, Some JW, Colaiezzi B, Do HTP, Rogers B. Accuracy and cost-effectiveness of the INDDEX24 Dietary Assessment Platform in Viet Nam. Br J Nutr. 2023 May 28;129(10):1751-1764. doi: 10.1017/S0007114522001507. Epub 2022 May 19. PMID 35587720
- [Background] Gibson RS, Charrondiere UR, Bell W. Measurement Errors in Dietary Assessment Using Self-Reported 24-Hour Recalls in Low-Income Countries and Strategies for Their Prevention. Adv Nutr. 2017 Nov 15;8(6):980-991. doi: 10.3945/an.117.016980. Print 2017 Nov. PMID 29141979
- [Background] Schutz Y. The basis of direct and indirect calorimetry and their potentials. Diabetes Metab Rev. 1995 Dec;11(4):383-408. doi: 10.1002/dmr.5610110406. No abstract available. PMID 8718497
- [Background] Murgatroyd PR, Shetty PS, Prentice AM. Techniques for the measurement of human energy expenditure: a practical guide. Int J Obes Relat Metab Disord. 1993 Oct;17(10):549-68. PMID 8242125
- [Background] Torun B. Energy requirements of children and adolescents. Public Health Nutr. 2005 Oct;8(7A):968-93. doi: 10.1079/phn2005791. PMID 16277815
- [Background] Burrows TL, Martin RJ, Collins CE. A systematic review of the validity of dietary assessment methods in children when compared with the method of doubly labeled water. J Am Diet Assoc. 2010 Oct;110(10):1501-10. doi: 10.1016/j.jada.2010.07.008. PMID 20869489
- [Background] Ukegbu PO. Energy intake, expenditure and body composition of adolescent boys and girls in public boarding secondary schools in Umuahia, Nigeria. J Biol Agric Healthc. 2012;2(8):33-9. Available from: https://iiste.org/Journals/index.php/JBAH/article/view/2860
- [Derived] Adegboyega MT, Amaeze CA, Uche CP, Ukegbu PO, Pontzer H. Study protocol for measuring energy needs and nutritional status of adolescent girls in Abia state, Nigeria: The nutrition and adolescence in rural Nigeria (NARN'ia) Study. PLoS One. 2025 Oct 7;20(10):e0333889. doi: 10.1371/journal.pone.0333889. eCollection 2025. PMID 41056327